CLINICAL TRIAL: NCT01116817
Title: Exploratory, Cross-sectional Study to Compare the Virologic Efficacy in Cerebrospinal Fluid (CSF) and Neurocognitive State in Patients Infected by HIV-1 Long-term Treatment (> 3 Years) With Lopinavir / Ritonavir Monotherapy
Brief Title: Study to Compare the Virologic Efficacy in Cerebrospinal Fluid (CSF) and Neurocognitive State in Patients Infected by HIV-1 Long-term Treatment (> 3 Years) With Lopinavir / Ritonavir Monotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCR-MONOKAL
Record Dates: First submitted 2010-04-30; First posted 2010-05-05 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: HIV
Keywords: Long-term Lopinavir/ritonavir monotherapy; neurocognitive performance; ultrasensitive CSF-viraemia
MeSH Terms: interventions — Spinal Puncture; Lopinavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LPV/r monotherapy 400/100 mg twice daily, orally administered (Experimental): LPV/r monotherapy 400/100 mg twice daily, orally administered
  Interventions: Drug: Lumbar puncture (Lopinavir/ritonavir monotherapy)
- Lumbar puncture (Active Comparator): LPV/r 400/100 mg twice daily + 2 NRTI, orally administered.
  Interventions: Drug: Lumbar puncture (HAART: Lopinavir/ritonavir + 2 NRTI)

INTERVENTIONS:
Drug: Lumbar puncture (Lopinavir/ritonavir monotherapy) — Lumbar puncture at week 0
  Other Names: NP
  Arms: LPV/r monotherapy 400/100 mg twice daily, orally administered
Drug: Lumbar puncture (HAART: Lopinavir/ritonavir + 2 NRTI) — Lumbar puncture at week 0
  Other Names: NP
  Arms: Lumbar puncture

SUMMARY:
The aim of this study is to describe and compare the percentage of patients infected by HIV-1 to maintain a complete virology suppression at the CSF (CSF CV 1 copy / mL) in patients with CV <50 copies / mL and treated with stable antiretroviral therapy for at least 3 years with LPV / r 400/100 mg twice daily + 2 NRTI.

DETAILED DESCRIPTION:
Combinations of antiretroviral for the management of HIV infection recommended by the main treatment guidelines include a combination of two nucleoside analogue reverse transcriptase (NRTI) with a non-nucleoside reverse transcriptase (NNRTI) or an inhibitor protease (IP) .1 However, NRTIs can inhibit mitochondrial DNA gamma polymerase, causing mitochondrial dysfunction, which in turn can result in related adverse effects such as peripheral neuropathy, pancreatitis, hepatitis, abnormal lipid profile or lipodystrophy. Therefore, it is advisable to design and search for therapeutic strategies to avoid prolonged exposure to NRTIs and their adverse events.

IP monotherapy as a strategy of simplification, after an induction period with standard triple therapy may be useful to minimize the risk of mitochondrial toxicity by NRTIs. Additionally, this strategy may be useful to improve treatment adherence, reduce costs and preserve future treatment options. In this sense, monotherapy with lopinavir / ritonavir (LPV / r) can be an effective option for the treatment of HIV-1 as a simplification strategy in routine clinical practice.3 OK04 study showed that in patients with sustained viral suppression simplified to monotherapy with LPV / r, rates of viral load <50 copies / mL were similar to that patients continuing on standard triple therapy.4, 5 However, the virological efficacy of this strategy in the CSF compartments has been questioned by some authors. Like most protease inhibitors, lopinavir has a poor penetration in CSF. Thus, despite the concentration of lopinavir in CSF usually exceed the inhibitory concentration (IC50) of wild strains of HIV, it is possible that some patients may present lopinavir concentrations insufficient to achieve sustained suppression of viral replication in that compartment. In this sense, according to results from a recent study, up to 10% of patients treated with lopinavir / ritonavir monotherapy may present detectable levels of viral load in CSF while maintaining a CV <50 copies / mL in plasma.9

On the other hand, about half of patients on antiretroviral therapy (HAART), despite achieving virologic control and the treatment is performed properly, have been neurocognitive dysfunction.10 This has been associated with multiple risk factors, including the presence of HIV in CSF.11 In fact, even though achieving undetectable viral load in plasma, up to 40% of patients on HAART show presence of virus in CSF.12 This also has been associated with a worse neurocognitive functioning. Therefore, the maximum control of viral replication is shown as a priority for the improvement of CNS dysfunction.

Based on the above, the objective of this study is to explore and evaluate the virological efficacy and safety at long-term neurocognitive level (> 3 years) of monotherapy with lopinavir / ritonavir as a strategy to simplify antiretroviral therapy in patients infected by HIV.

ELIGIBILITY:
Inclusion Criteria:

Experimental group:

1. Patients having a diagnosis of HIV infection, on stable treatment at least 3 years with LPV/r monotherapy, the inclusion of patients with at least 2 years will be permitted if it is not possible to include the expected number of patients.
2. Initiating monotherapy with lopinavir / ritonavir maintaining values of plasma HIV-1 RNA undetectable (cv <50 copies / mL).
3. Maintain complete virologic suppression (CV <50 copies / ml) in plasma for at least 3 years in treatment with LPV / r monotherapy. (Or 2 years, if not complied with the expected number of patients with at least 3 years with LPV / r monotherapy).
4. Good adherence to treatment (> 90%).
5. Signing of informed consent.

Control group:

1. Patients having a diagnosis of HIV infection, on stable treatment at least 3 years with LPV/r 400/100 mg twice a day + 2 ITIAN, the inclusion of patients with at least 2 years will be permitted if it is not possible to include the expected number of patients.
2. Maintain complete virologic suppression (CV <50 copies / ml) in plasma for at least 3 years in treatment with LPV / r monotherapy. (Or 2 years, if not complied with the expected number of patients with at least 3 years with LPV / r 400/100 mg 2 twice a day + 2 ITIAN).
3. Patients that can be put into pairs with the experimental ones following these characteristics: age, sex, presence of previous virologic failures, nadir CD4 + T lymphocytes and viral load <50 copies / mL time prior to inclusion in the study. Patients having a diagnosis of HIV.
4. Good adherence to treatment (> 90%).
5. Signing of informed consent.

Exclusion Criteria:

1. Vaccine administration, acute or chronic uncontrolled infection in the 2 months prior to the inclusion or medical assessment which in the opinion of the investigator, might compromise the results of the study.
2. Pregnancy or breastfeeding.
3. Therapies that include interferon, interleukin-2, cytotoxic chemotherapy or immunosuppressant at baseline.
4. Do not sign the informed consent.
5. Existence of any contraindication to the performance of lumbar puncture.
6. Presence of psychiatric disorders or being in psychopharmacological treatment.
7. Active alcohol consumption (> 50 g / day) or illicit drugs.
8. Existence current or past opportunistic infection involving CNS functioning alteration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Ultrasensitive HIV-1 RNA in CSF | week 0

SECONDARY OUTCOMES:
CD4 cell count | week 0
Plasmatic HIV-1 Viral load | week 0
Plasmatic and CSF trough-LPV concentration | weeks 0
Neurocognitive alteration, present when there is a diagnosis of any neurocognitive disorders associated with HIV (HAND). | week 0
Overall deficit ratio (GDS) | week 0
  Calculating a value of overall neurocognitive functioning, based on an evaluation of 7 representative areas in HIV infection (attention / working memory, speed of information processing, verbal memory, learning, verbal fluency.
Adverse events | week 0

CONTACTS AND LOCATIONS:
Locations (1):
- Germans Trias i Pujol Hospital, Badalona, Barcelona, Spain